CLINICAL TRIAL: NCT04673708
Title: Using H - Test to Identify the Sexual Orientation and Applying the Test in Medical and Forensic Fields
Brief Title: H - Test Usage in Identification of Sexual Orientation Among People.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hashim Talib Hashim, Clinical researcher, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: H98
Record Dates: First submitted 2020-11-28; First posted 2020-12-17 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Sexual Behavior; Sexual Orientation Conflict Disorder; Sexual Arousal Disorder; Sexual Orientation; Sexual; Orientation, Relationship Disorder
MeSH Terms: conditions — Sexual Behavior; Sexual Dysfunctions, Psychological; Coitus; Orientation, Spatial

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hashim Talib Hashim (Other): It is a video with +18 different contents to know the effect of much video than the others.
  Interventions: Diagnostic Test: H - Test
- Mustafa Ahmed Ramadhan (Experimental): Is is an assessment of the vital signs among the participants and the change with the showing of videos.
  Interventions: Diagnostic Test: H - Test

INTERVENTIONS:
Diagnostic Test: H - Test — Showing different videos for a sexual stimulus and monitor the vitals of each participants to measure any changes can occur with each video.
  Other Names: Sexual desire test; Sexual health test

SUMMARY:
Using of H - test in identifying the sexual behavior of the human.

DETAILED DESCRIPTION:
The test using videos and in the same time watching the vital signs of the participant to identify any changes in them align with the vides.

These videos contain +18 contents that can excite them and make them sexually active. So we can determine with type of vides that more excited to the human and select his or her sexual behavior type.

ELIGIBILITY:
Inclusion Criteria:

* All the people can be included

Exclusion Criteria:

* Have a psychological disorder
* Have a sexual disorder

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-26 (Actual)

PRIMARY OUTCOMES:
An observatory stimulation test of sexual orientation (Straight, gay, lesbian, bisexual) by using videos stimulation | 1 week
  Using the test to arouse the sexual state among the participants by using sexual videos either for gays or straights, that can stimulate them sexually while monitoring their vitals to see the changes that can occur with each videos and the most effective video will be considered as a sufficient stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Talib Manea, MD, Study Chair — University of Thi-Qar
Locations (1):
- No name, Nasiriyah, Thi Qar, Iraq

IPD SHARING:
Plan to Share IPD: Yes
No personal data will be shared with others except the data used to state the study measures.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: They will be available in three months and for six months.
Access Criteria: They will shared on drive